CLINICAL TRIAL: NCT07197476
Title: Adolescent Injury: Intervening to Prevent Posttraumatic Stress and Substance Use Outcomes
Brief Title: Adolescent Stress and Substance Intervention Subsequent to Trauma
Acronym: ASSIST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DA062071 (NIH); 1R21DA062071 (NIH)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: PTSD; Substance Use Disorder (SUD); Acute Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Develop and Pilot Test ASSIST Video Intervention (Experimental): The investigators will develop and pilot test the Adolescent Stress and Substance Intervention Subsequent to Trauma (ASSIST) video intervention that builds upon ACS-COT guidelines to improve mental health care during and after hospitalization for traumatic injury. The ASSIST video intervention is a simple, cost-effective, and scalable tool that may be easily integrated into usual care settings to address posttraumatic symptoms and decrease risk of subsequent substance use following discharge.
  Interventions: Behavioral: ASSIST Video Intervention

INTERVENTIONS:
Behavioral: ASSIST Video Intervention — Video intervention for participants: adolescent trauma patient-parent dyads.

SUMMARY:
The long-term goal of this study is to address the adoption of the new trauma center requirement to establish best practices of screening for acute stress with an intervention to prevent both adolescent PTSD and substance use. The investigators will develop, refine, and pilot test the Adolescent Stress and Substance Intervention Subsequent to Trauma (ASSIST) video interventions that build upon the American College of Surgeons Committee on Trauma guidelines to improve mental health care during and after hospitalization for traumatic injury. The aims are:

PHASE I - Primary Aim 1: To develop and refine two ASSIST video interventions for adolescents and parents admitted to a level 1 pediatric trauma center.

PHASE II

* Primary Aim 2a: To evaluate the feasibility, acceptability and implementation potential of the ASSIST video interventions.
* Primary Aim 2b: Develop the ASSIST implementation protocol using a national advisory panel of pediatric trauma center leaders.

Participants in PHASE 1:

Parent and child duo:

* Review storyboards for the video interventions
* Participate in qualitative interviews at hospital admission and 1 month following discharge

Pediatric trauma center clinical staff members:

- Complete qualitative interviews

Participants in PHASE II:

Parent and child duo:

* Shown their own video interventions
* Complete assessments at admission and 1-, 2-, 3- months after discharge

ELIGIBILITY:
Inclusion Criteria for Youth:

* Must be 12-17 years
* Fluent in English or Spanish
* Able to provide informed assent
* Have a parent able to provide informed consent

Inclusion Criteria for Parents:

* Live with an admitted pediatric trauma patient
* Fluent in English or Spanish
* Able to provide informed consent

Exclusion Criteria:

* Prisoner or in police custody
* Involvement with child protective services
* Admitted due to suicide attempt or non-suicidal self-injury
* Any acute condition that would preclude provision of informed consent or assent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To develop and refine two ASSIST video interventions for adolescents and parents admitted to a level 1 pediatric trauma center. | 30 days
  Elicit feedback from content experts to further refine initial ASSIST video interventions. Conduct qualitative interviews with 15-20 parents and adolescents (12-17 years) to assess perceived usefulness of, and satisfaction with, intervention content as well as elicit feedback on areas for future refinement.
  Conduct qualitative interviews with 9-12 key stakeholders in the fields of pediatric trauma care to assess clinical concerns/strategies as well as implementation barriers/facilitators.
To evaluate the feasibility, acceptability, and implementation potential of the ASSIST video interventions. | 3 months
  Examine the feasibility and acceptability of the ASSIST videos, over a 3-month period, as measured by rates of enrollment and retention, interest/satisfaction, knowledge regarding mental health symptoms/substance use, incidence (quantity/frequency) of substance use, self-efficacy in having discussions about mental health symptoms/ substance use, self-efficacy around connecting participant's child to mental health and/or addiction resources, and (when appropriate) engagement with a provider for mental health and/or addiction care.
Develop the ASSIST implementation protocol | 3 months
  Develop the ASSIST implementation protocol using a national advisory panel of pediatric trauma center leaders. Using an expert panel from the national cohort of pediatric trauma centers the investigators have worked with in a previous implementation trial, and pilot data from the investigators' institution, an implementation protocol will be developed that will be tested in a subsequent fully powered R01 hybrid implementation-efficacy trial.